CLINICAL TRIAL: NCT03497494
Title: Analysis the Related Factors of Bariatric Surgery on Gastroesophageal Reflux Disease and Its Prevention and Treatment: a Prospective, Multicenter and Randomized Controlled Study
Brief Title: the Related Factors of Bariatric Surgery on Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Jingge Yang, Director of bariatric surgery, First Affiliated Hospital of Jinan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FirstJinanU20180120
Record Dates: First submitted 2018-03-15; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Gastroesophageal Reflux; Bariatric Surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: All patients enrolled in this study underwent laparoscopic sleeve gastrectomy. According to the starting point of resection to pylorus distance and whether to the strengthen suture of esophageal hole, the cases were randomly divided into 6 groups:
  G1: 2 cm away from the pylorus edge, without hiatal suture; G2: 4 cm away from the pylorus edge, without hiatal suture; G3: 6 cm away from the pylorus edge, without hiatal suture; G4: 2 cm away from the pylorus edge, with hiatal suture G5: 4 cm away from the pylorus edge, with hiatal suture; G6: 6 cm away from the pylorus edge, with hiatal suture;
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without hiatal suture (Active Comparator): the different distance of pylorus without hiatal suture
  Interventions: Procedure: 2 cm away from the pylorus edge; Procedure: 4 cm away from the pylorus edge; Procedure: 6 cm away from the pylorus edge; Procedure: LRYGB
- With hiatal suture (Active Comparator): the different distance of pylorus without hiatal suture
  Interventions: Procedure: 2 cm away from the pylorus edge; Procedure: 4 cm away from the pylorus edge; Procedure: 6 cm away from the pylorus edge

INTERVENTIONS:
Procedure: 2 cm away from the pylorus edge — 2 cm away from the pylorus edge
Procedure: 4 cm away from the pylorus edge — 4 cm away from the pylorus edge
Procedure: 6 cm away from the pylorus edge — 6 cm away from the pylorus edge
Procedure: LRYGB — laparoscopic Roux-en-Y gastric bypass
  Other Names: laparoscopic Roux-en-Y gastric bypass
  Arms: Without hiatal suture

SUMMARY:
Obesity and related metabolic diseases have become a chronic disease that is a threat to human health. Bariatric surgery can effectively and long-term reduce excess body weight and relieve related metabolic diseases, including type 2 diabetes. Laparoscopic gastric bypass surgery and laparoscopic sleeve gastrectomy are commonly used in bariatric surgery. Laparoscopic sleeve gastrectomy due to simple operation, good weight loss, and metabolic disease control effect, which is more widely used. However, there are several studies that show an increased chance of gastroesophageal reflux disease after laparoscopic sleeve gastrectomy. Long-term gastroesophageal reflux may lead to Barrett's esophagus or esophageal cancer. Nowadays, the cause of gastroesophageal reflux disease after sleeve gastrectomy is not clear and precautionary measures are not precise.

In this study, prospective randomized controlled trials were conducted to explore the possible causes of gastroesophageal reflux after sleeve gastrectomy and to explore ways to prevent gastroesophageal reflux disease after sleeve gastrectomy.

DETAILED DESCRIPTION:
With the social development and changes in the lifestyle, the incidence of obesity and type 2diabetes is rapidly increasing. In 2010, the global incidence of type 2 diabetes was 8.3% in adults, 11.6% in China and 50.1% in China. In overweight and obese people, the prevalence of type 2 diabetes also increased significantly, and the prevalence of type 2diabetes in those people with BMI> 30 reached 18.5-23%. Diabetes-induced cardiovascular and cerebrovascular diseases, renal insufficiency and other complications, seriously affecting the quality of life of the patients, endangering the safety of life, the treatment of type 2 diabetes and related complications to public health expenditure has brought tremendous pressure.

Traditional medical methods are difficult to achieve long-term and effective control of type 2 diabetes. Surgery has been shown to achieve 75-95% long-term relief of obesity in patients. Roux-en-Y gastric bypass (Roux-en-Y gastric bypass, RYGB) and laparoscopic sleeve gastrectomy are most commonly used. Among them, laparoscopic sleeve gastrectomy is relatively simple, low incidence of complications, lower operating costs, and gradually become the most important surgical methods of weight loss and metabolic disease surgery. Numerous clinical studies are shown that sleeve gastrectomy in patients with type 2 diabetes has the same therapeutic effect as gastric bypass with a complete remission rate of 70-90% for T2DM.

For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, participants can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In China, the BMI less than 45 is majorities.

According to the previous survey in 2012, the newly diagnosed diabetes patients in China constituted more than half of all diabetic patients. Since laparoscopic sleeve gastrectomy is relatively simple, so sleeve gastrectomy is easier to popularize in China and has wide application prospect.

As an invasive treatment, laparoscopic sleeve gastrectomy also presents opportunities of surgery-related complications, including gastric leak (0.5-1%), stenosis (0.1-0.5%), bleeding (about 0.5%), and gastroesophageal reflux disease (GERD). Gastroesophageal reflux disease is a most common upper gastrointestinal disease, numerous clinical studies shown that the incidence of GERD in western populations are 10-20%, while obese people are around 37-72%, if abdominal fat accumulation more obvious, the incidence of GERD will become higher. In China, there is still no relevant data. Gastric bypass surgery has a clear effect on the treatment of GERD, and the relationship between sleeve gastrectomy and GERD is still controversial. Some studies have shown that sleeve gastrectomy did not increase the incidence of postoperative GERD, while another study showed that the incidence of GERD after sleeve gastrectomy increased significantly. In addition, no studies have revealed the reasons for the occurrence of GERD after sleeve gastrectomy and no study showed how to prevent the occurrence of GERD after sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, you can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In our country, the BMI less than 45 is majorities.

Exclusion Criteria:

* BMI<27.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
GERD-Health Related Quality of Life Questionnaire | 1 year
  Total Score: Calculated by summing the individual scores to questions 1-15.
  * Greatest possible score (worst symptoms) = 75
  * Lowest possible score (no symptoms) = 0 Heartburn Score: Calculated by summing the individual scores to questions 1-6 .
  * Worst heartburn symptoms = 30
  * No heartburn symptoms = 0
  * Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination. 2 Regurgitation Score: Calculated by summing the individual scores to questions 10-15.
  * Worst regurgitation symptoms = 30
  * No regurgitation symptoms = 0
  * Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

SECONDARY OUTCOMES:
preoperative and postoperative of abdominal ultrasound to examine the abdominal fat thickness | 1 year
  abdominal fat thickness in centimeter
Preoperative and postoperative BMI | 1 year
  The patient's weight and height will be combined to report BMI in kg/m^2
Preoperative and postoperative waist circumference | 1 year
  waist circumference in centimeter
Preoperative and postoperative abdominal circumference | 1 year
  abdominal circumference in centimeter
Preoperative and postoperative chest circumference | 1 year
  chest circumference in centimeter
Preoperative and postoperative neck circumference | 1 year
  neck circumference in centimeter
Preoperative and postoperative bone mineral density | 1 year
  bone mineral density in percentage
Preoperative and postoperative body fat measured | 1 year
  body fat measured in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- The frist affiliated hospital of Jinan University, Guangzhou, Guangdong, China